CLINICAL TRIAL: NCT00474981
Title: Impact of the Integrated Management of Neonatal and Childhood Illness Strategy on Neonatal and Infant Mortality in Haryana, India
Brief Title: Impact of the Integrated Management of Neonatal and Childhood Illness Strategy on Neonatal and Infant Mortality
Acronym: IMNCI-India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Society for Applied Studies (Other)
Collaborators: World Health Organization (Other); United Nations (Other); The Research Council of Norway (Other); Society for Essential Health Action and Training, New Delhi - Year 3 onwards (Unknown)
Responsible Party: Principal Investigator, NBhandari, Director, Society for Applied Studies
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: C6-181-505
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-04

CONDITIONS: Mortality
Keywords: neonatal mortality; infant mortality; newborn caring practices
MeSH Terms: conditions — Infant Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): IMNCI
  Interventions: Behavioral: IMNCI
- 2 (No Intervention): Control

INTERVENTIONS:
Behavioral: IMNCI — Implementation of IMNCI in the intervention sites
  Arms: 1

SUMMARY:
This study is a cluster-randomized trial being conducted in the state of Haryana in North India. Eighteen geographical areas served by Primary Health Centres (PHCs) have been randomized to intervention or comparison areas. In the intervention areas, all physicians, health workers and ICDS workers are being trained in the IMNCI. Each of these clusters has an approximate population of 30,000.

The IMNCI intervention includes three main components:

1. improvement in the case management skills of health staff
2. improvement in the overall health system to support its performance, and
3. improvement in family and community health care practices which include:

   * prevention and management of hypothermia
   * early initiation of breastfeeding and exclusive breastfeeding
   * community-based care of low birth weight infants
   * improved care-seeking for neonatal infections

The primary outcome measures of the study are neonatal and infant mortality. The study will also collect information on cause-specific neonatal mortality, ascertained using a standardized previously validated verbal autopsy instrument administered by trained, skilled health workers. All the other outcomes (including initiation of breastfeeding within 1 hour of birth; Exclusive breastfeeding at 4 weeks of age; Proportion of neonates identified to be sick by caregivers who sought care) are secondary outcomes.

The effectiveness of this comprehensive intervention will be measured by comparing the primary and secondary outcome measures in the intervention and comparison clusters, controlling for any baseline differences such as the predefined outcomes and/or socioeconomic status and demography.

The project will serve as a guide to the Government of India of how to best implement the IMNCI strategy and measure its impact.

DETAILED DESCRIPTION:
OBJECTIVES

The primary objective of this study is to determine the effectiveness of delivering community and facility based newborn interventions as part of the IMNCI strategy:

* in reducing (i) neonatal mortality beyond the first 24 hours of birth, i.e. from 1-28 days of age and (ii) overall neonatal mortality, i.e. from birth to 28 days of age, in the communities receiving the intervention [based on a cohort of infants born to women identified through pregnancy surveillance]
* in reducing (i) neonatal mortality beyond the first 24 hours of life (day 1-28) and (ii) overall neonatal mortality (birth to 28 days of age) in the population of newborns more likely to have greater impact from the intervention, i.e. those born at home and available in the study area within 7 days of birth [based on a cohort of infants born at home and available in the study area within 7 days of birth]
* in reducing infant mortality (from birth to 365 days of age) in the intervention communities [based on a cohort of infants born to women identified through pregnancy surveillance]

The secondary objectives of the study are to determine the effectiveness of delivering community and facility based newborn interventions as part of the IMNCI strategy:

- in improving newborn care practices in households.

SAMPLE SIZE ESTIMATES

Sample size estimates were revised subsequent to the expansion of the primary objectives and completion of one year of surveillance.

Cohort identified through pregnancy surveillance: The average neonatal mortality rate in the 18 sites in the first year of the study was 42 (range 31-52 ) in the cohort of infants born to women identified through pregnancy surveillance .The neonatal mortality rate beyond the first 24 hours of birth in the same cohort was 24 (range 19-31). We estimated that on an average 3700 neonates per cluster would be enrolled over the study enrollment period of 27 months after taking into account 10% attrition, to detect 20% difference in mortality with 80% power and 95% confidence level.

Population more likely to have greater impact from the intervention: The average neonatal mortality rate in the target population of newborns who are more likely to benefit from the intervention i.e. those born at home and available in study area within 7 days of birth was 36 (range 19-43). The mortality beyond the first 24 hours of birth in the same cohort was 22 (range 13-25). On an average 2000 neonates per cluster would be enrolled over the study enrollment period of 27 months. This would enable us to detect 25% difference in mortality with 80% power and 95% confidence level.

To summarise, 27 months of enrollment will give 80% or more power to detect:

In the pregnancy cohort:

* 20% or greater reduction in neonatal mortality.
* 20% in the mortality of neonates beyond first 24 hours of birth.

In the population more likely to have greater impact (i.e. those born at home and available in the study area within 7 days of birth):

* 25% or greater reduction in mortality from birth to 28 days
* 25% or greater reduction in the neonatal mortality beyond first 24 hours of birth.

The sample size has also been estimated for process evaluation outcomes through observations at health facilities (quality of care at health facilities) and exit interviews (knowledge and skills of mothers on home care of illness). Our guesstimates of the proportions in the control group are based on experience of working in the area. The number of clusters was taken as 9 per group based on sample size calculations for mortality discussed above. The table below shows that 50 observations and 50 exit interviews per cluster (i.e. 450 observations and exit interviews each in the intervention clusters and 450 in the control clusters i.e. a total of 1800) would be adequate to detect a 20% absolute increase in the outcome with 90% power.

THE INTERVENTION

The intervention was designed following the guidelines developed by the Government of India in collaboration with the WHO and UNICEF (2). The intervention includes three main components:

1. Improving the case management skills of health staff: Qualified physicians, supervisors and other health workers in the intervention sites along with anganwadi workers will be trained in IMNCI through an 8 day course. A set of information meetings will be designed for traditional birth attendants registered medical practitioners and qualified physicians working in the private sector. The training will be completed by a visit to the trainee at his/her work place within 1 month of the course to review the performance, correct any problems and support the use of the skills taught during the course.
2. Strengthening of health systems.

   As part of its collaboration with the project, efforts will be undertaken by the District Medical Officer's team to implement the following health systems improvements with a focus on the intervention areas:

   Availability of drugs and supplies needed for IMNCI: In order to ensure availability of essential IMNCI drugs and supplies a checklist will be prepared and displayed in the health facility. This list will be used as a checklist during Supervisory Visits.

   Improving referral pathways and services: Facilities will keep records of cases attended, cases referred and problems reviewed in supervisory visits and review meetings between the program in charge from the local health team and different categories of health workers.

   Supervisory Visits: Both scheduled and unscheduled visits will be conducted by supervisors (belonging to the local heath system and those provided through this project) trained in IMNCI. Supervisors will review the availability of facility supports and drugs to implement IMNCI, as well as health workers performance, and provide feedback and help problem-solving.
3. Improvement in family and community practices.

The aim of this component of the IMNCI strategy is to initiate, reinforce and sustain the key family practices for child survival, growth and development. Practices that are of particular importance for newborn health (early initiation of breastfeeding and avoidance of pre-lacteal feeds; keeping the baby warm, avoiding early bathing, cord hygiene, care seeking for danger signs and special attention for LBW newborns) will be promoted in addition to the standard IMCI key practices (3).

OUTCOME ASCERTAINMENT

One field worker will be allocated 2000 to 3000 households and will keep his/her area under surveillance to identify pregnant women. For all pregnancies identified, visits will be made to the household on a day coinciding with infant age ~1 month to document the outcome of pregnancy. Subsequent visits will be made at infant age 3, 6, 9 and 12 months to record the vital status of the infant.

PROCESS EVALUATION ACTIVITIES

These will be conducted by a 6 member team both in the intervention and control clusters and will essentially focus on activities that ascertain how well the intervention is being implemented. The evaluation will be conducted in a small subsample of the various activities in each of the 18 clusters and will include the following:

* Observations of health care providers, consultations with caregivers of infants aged < 29 days and infants between 1 to 11 months of age
* Exit interviews with mothers who have recently visited a health care provider for treatment of illness in an infant aged < 29 days and infants between 1 to 11 months of age.
* Interviews with caregivers/mothers with a young infant who were home visited recently by a health worker

DATA MANAGEMENT

Forms filled in the field will be manually self-checked for missing information, data range and consistency by the person filling the form. A double data entry system will be used followed by validation and merging of the double entered cleaned data.

ANALYSIS

Socioeconomic, environmental and demographic characteristics of the intervention and control clusters will be examined for group comparability. Any significant differences will be controlled for during data analysis. The potential confounders on which data will be collected at baseline include:

* Distance from the nearest government outpatient facility
* Distance from the nearest private outpatient facility
* Distance from the nearest government inpatient facility
* Distance from the nearest private inpatient facility
* Density of private providers
* Density of qualified private providers
* Number of private practitioners used for care of infants

The frequencies of the main study variables will be examined to assess the distribution of data. If the data are not normally distributed, decisions about the need for data transformation and the appropriateness of statistical tests will be made.

Efficacy evaluation will be done by comparing the primary and secondary outcome measures in the intervention and control clusters, controlling for any socioeconomic, environmental or demographic differences.

To account for the clustered nature of the data, techniques such as Generalized Estimating Equation and multi-level modelling will be used.

Data analysis will be carried out using Stata, Version 8.2.

REFERENCES

1. Smith PG, Morrow RH. Field trials of health interventions in developing countries: a toolbox. London: Macmillan Education, 1996
2. Government of India. Operational Guidelines for Implementation of Integrated Management of Neonatal and Childhood Illness (IMNCI). Ministry of Health Family Welfare: New Delhi, 2006.
3. World Health Organization. Integrated Management of Childhood Illness. Geneva: World Health Organization, 1997 (WHO/CHD/97.3E).

ELIGIBILITY:
Inclusion Criteria:

* All births

Exclusion Criteria:

* None

Ages: 1 Minute to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66600 (Actual)
Dates: Start 2006-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Post day 1 Neonatal mortality (birth to 28 days of age) in the communities receiving the intervention(cohort of infants born to women identified through pregnancy surveillance) | Over 30 Months
Neonatal mortality (from birth to 28 days of age) in the cohort identified through pregnancy surveillance | Over 30 Months
Post day 1 neonatal mortality (1 to 28 days of age) in the population of newborns who are more likely to have greater impact from the intervention i.e. those born at home and available in the study area within 7 days of birth | 30 months
Neonatal mortality (from birth to 28 days of age) in the population more likely to benefit from the intervention | 30 months
Infant mortality (birth to 365 days) in the communities receiving the intervention. | 30 months

SECONDARY OUTCOMES:
Population coverage of key behaviours and interventions | Over 30 Months
Process of intervention delivery in a randomly selected subsample of activities | Over 30 Months

CONTACTS AND LOCATIONS:
Overall Officials: Nita Bhandari, MD, PhD, Principal Investigator — Society for Applied Studies
Locations (1):
- Society for Applied Studies, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Result] Bhandari N, Mazumder S, Taneja S, Sommerfelt H, Strand TA; IMNCI Evaluation Study Group. Effect of implementation of Integrated Management of Neonatal and Childhood Illness (IMNCI) programme on neonatal and infant mortality: cluster randomised controlled trial. BMJ. 2012 Mar 21;344:e1634. doi: 10.1136/bmj.e1634. PMID 22438367
- [Derived] Chowdhury R, Taneja S, Mazumder S, Bhandari N, Strand TA. Gender differences in infant survival: a secondary data analysis in rural North India. BMJ Open. 2017 Aug 11;7(8):e014179. doi: 10.1136/bmjopen-2016-014179. PMID 28801386
- [Derived] Taneja S, Bahl S, Mazumder S, Martines J, Bhandari N, Bhan MK. Impact on inequities in health indicators: Effect of implementing the integrated management of neonatal and childhood illness programme in Haryana, India. J Glob Health. 2015 Jun;5(1):010401. doi: 10.7189/jogh.05.010401. PMID 25674350
- [Derived] Mazumder S, Taneja S, Bahl R, Mohan P, Strand TA, Sommerfelt H, Kirkwood BR, Goyal N, Van Den Hombergh H, Martines J, Bhandari N; Integrated Management of Neonatal and Childhood Illness Evaluation Study Group. Effect of implementation of integrated management of neonatal and childhood illness programme on treatment seeking practices for morbidities in infants: cluster randomised trial. BMJ. 2014 Aug 29;349:g4988. doi: 10.1136/bmj.g4988. PMID 25172514